CLINICAL TRIAL: NCT06361316
Title: Efficacy and Safety of Irinotecan Liposome Injection Combined With Oxaliplatin and Tegafur (NASOX) in Adjuvant Chemotherapy for Pancreatic Cancer
Brief Title: Irinotecan Liposome Combined With Oxaliplatin and Tegafur as Adjuvant Therapy for Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuirong Jiang (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Kuirong Jiang, archiater, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PC-JS01
Record Dates: First submitted 2024-03-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Pancreatic Cancer; Adjuvant Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Irinotecan liposome injection+ Oxaliplatin +Tegafur (Experimental): Oxaliplatin: 60mg/m2, d1, ivgtt, 2h; Repeat every 15 days; Irinotecan liposomes: 50mg/m2, d1, ivgtt, 90min; Repeat every 15 days; Tegafur: 40-60mg, BID, po, d1-d10, repeat every 15 days; 30 days as one cycle, 6 treatment cycles.
  Interventions: Drug: Irinotecan liposome injection

INTERVENTIONS:
Drug: Irinotecan liposome injection — Postoperative adjuvant therapy
  Other Names: oxaliplatin; Tegafur

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of irinotecan liposome injection in combined with oxaliplatin plus tegafur (NASOX) for postoperative adjuvant chemotherapy for pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. ECOG performance status 0 or 1.
2. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1).
3. ECOG performance status 0 or 1.
4. Life expectancy of greater than or equal to 6 months.
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Patients who cannot eat orally and have gastric emptying disorder after surgery;
2. Patients with moderate diarrhea: diarrhea ≥4 times per day; the moderate and severe effluents from stoma increased; Or diarrhea that limits activities of daily living;
3. Patients who cannot eat orally and have gastric emptying disorder after surgery;
4. Patients who cannot eat orally and have gastric emptying disorder after surgery;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival, DFS | baseline up to approximately 21.6 months.
  the time from the start of randomization (or the start of treatment in a one-arm trial) to the recurrence of disease or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Adverse events (aes) were determined and graded according to NCI-CTCAE version 5.0, and evaluated by the overall incidence of AE, the incidence of AE grade 3 or above, and the incidence of SAE | baseline up to approximately 7 months.
  Hematologic and non-hematologic adverse events during adjuvant therapy (according to NCI-CTCAE5.0);
Overall Survival, OS | baseline up to approximately55 months.
  the time from the start of randomization (or the start of treatment in a one-arm trial) to death from any cause.
Quality of life, QOL | baseline up to approximately 55 months.
  It reflects the ability of human activities to improve the survival level and survival chances, evaluated according to EORTC Quality of life measurement scale QLQ-C30 V3.0 assessment.
The results were presented in terms of the proportion of patients who completed 6 months of chemotherapy | baseline up to approximately 7 months.
  The results were presented in terms of the proportion of patients who completed 6 months of chemotherapy
he results were presented in terms of the proportion of patients who were replaced with 5-FU/LV due to Tegafur intolerance | baseline up to approximately 7 months.
  The results were presented in terms of the proportion of patients who completed 6 months of chemotherapy and the proportion of patients who were replaced with 5-FU/LV due to Tegafur intolerance

CONTACTS AND LOCATIONS:
Overall Officials: KuiRong Jiang, archiater, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- FirstNanjingMU, Nanjing, Jiangsu, China